CLINICAL TRIAL: NCT00113802
Title: A Phase II, Single-Arm Trial of Epratuzumab, an Anti-CD22 Humanized Antibody, in Patients With Waldenstrom's Macroglobulinemia
Brief Title: Study of Epratuzumab (hLL2) in Patients With Waldenstrom's Macroglobulinemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low accrual
Sponsor: Gilead Sciences (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM-T-hLL2-18-US
Record Dates: First submitted 2005-06-10; First posted 2005-06-13 (Estimated); Last update posted 2021-08-19 (Actual); Status verified 2008-02

CONDITIONS: Waldenstrom Macroglobulinemia
Keywords: Epratuzumab (hLL2- anti-CD22 humanized antibody); Waldenstrom's Macroglobulinemia; Waldenstrom Macroglobulinemia; Hematologic Disease; Hematologic Diseases; Paraproteinemias; Vascular Hemostatic Disorders; Lymphoproliferative Disorders
MeSH Terms: conditions — Waldenstrom Macroglobulinemia; Hematologic Diseases; Paraproteinemias; Hemostatic Disorders; Lymphoproliferative Disorders | interventions — epratuzumab

INTERVENTIONS:
Drug: Epratuzumab (hLL2- anti-CD22 humanized antibody)

SUMMARY:
The purpose of this study is to determine whether epratuzumab provides effective therapy in Waldenström's Macroglobulinemia (WM).

DETAILED DESCRIPTION:
This multi-center, single-arm study of epratuzumab is in patients with Waldenström's Macroglobulinemia (WM) who failed chemotherapy. After baseline evaluations, patients receive epratuzumab infused over approximately 30-60 minutes at 360 mg/m2, administered once weekly for 4 consecutive weeks (days 1, 8, 15, 22). Post-treatment evaluations occur on the day of the last infusion, then at 6 and 12 weeks. Patients without progression of disease continue long-term follow up until disease progression or for at least 5 years, with evaluations every 3 months for 2 years, then semi-annually. Otherwise, follow-up is only required until resolution of any treatment related abnormalities.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of Waldenström's Macroglobulinemia using criteria proposed at 2nd International Workshop on WM, Athens, Greece, 2002.
* Measurable disease, defined as serum monoclonal IgM protein ≥1000 mg/dL by electrophoresis.
* Lymphoplasmacytic infiltration of the bone marrow >10% involvement.
* Failed at least one, but no more than 3, regimen(s) of prior therapy.

(Please consult with study site for full eligibility criteria)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31
Dates: Start 2004-08; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Serum measurements of IgM will be the primary determination of efficacy.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Weill Medical College of Cornell/ New York Presbyterian Hospital, New York, New York
  - Columbia University College of Physicans & Surgeons, New York, New York